CLINICAL TRIAL: NCT00959712
Title: Computer Agents to Promote Walking in Older Adults With Low Health Literacy
Brief Title: Computer Agents to Promote Walking in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Northeastern University (Other); Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01AG028668 (NIH)
Record Dates: First submitted 2009-08-14; First posted 2009-08-17 (Estimated); Last update posted 2023-06-29 (Actual); Status verified 2011-11

CONDITIONS: Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Subjects are given a pedometer and step count log in which to record their daily step counts for 1 year.
- ECA Interaction (Active Comparator): Subjects are given pedometers and step count logs in which to record their daily steps for 1 year. Subjects are also given a tablet computer and instructed to interact with the ECA (Embodied Conversational Agent) "Tanya" every day for 2 months.
  Interventions: Behavioral: ECA Interaction

INTERVENTIONS:
Behavioral: ECA Interaction — The technology uses a computer character (Embodied Conversational Agent (ECA)) that simulates face-to-face conversation. The ECA talks to the patient and the patient responds by tapping a touch-screen.
  Arms: ECA Interaction

SUMMARY:
This proposal is a randomized control trial using innovative interactive health technologies to promote and sustain walking behavior among elderly patients. The technology uses an Embodied Conversational Agent (ECA), a computer character that simulates face-to-face conversation. The trial will be block randomized by literacy status and include an intensive two-month, daily contact intervention via a Tablet PC ECA in the subject's home, an automated telephone program, and then an in-clinic, kiosk-based ECA for an additional 10 months, to promote maintenance of walking behavior. The study will occur in 2 phases, a pilot phase in which 20 subjects will be enrolled for the purpose of pre- testing the intervention and all data collection instruments, and a main study phase in which an additional 264 subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. 65 years old or greater
2. English-speaking
3. Actively being cared for by a primary care provider at Boston Medical Center

Exclusion Criteria:

1. Non-ambulatory
2. Any medical condition or disorder that would limit participation in moderate intensity physical activity (such as sustained walking), including life-threatening disorders, myocardial ischemia, complex cardiac arrhythmias or significant left ventricular dysfunction, and major functional disabilities relating to gait or balance
3. Medications that would compromise patient's ability to participate
4. Had more than 2 falls in the past year (i.e. fall risk)
5. Moderate to severe dementia
6. Severe depression
7. Currently exercising, i.e., engaged regularly in moderate-intensity or more vigorous physical activity 3 or more days per week for at least 20 minutes per day

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 263 (Actual)
Dates: Start 2008-10; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Increase in physical activity (measured as step counts from pedometer) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca A Silliman, MD, PhD, Principal Investigator — Boston University